CLINICAL TRIAL: NCT03889938
Title: Serum Level of Bioactive Mediators and Urinary Biopyrins in Psoriasis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Mahrous, Principal investigator, Assiut University
Other Study IDs: BMP
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serum and urinary assessment — Assess bioactive lipid mediators in blood and biopyrins in urine

SUMMARY:
1. Assess the level of lipid mediators in patients with psoriasis
2. Assess the urinary level of biopyrins as New marker of oxidative stress in patients with psoriasis
3. Correlate the serum level of bioactive lipid mediators and urinary level of biopyrins with Psoriasis Area and Severity Index

DETAILED DESCRIPTION:
Psoriasis is acommon immune mediated inflammatory skin disorder of complex pathomechanisms which is generically conditioned and influenced by environmental factors

ELIGIBILITY:
Inclusion Criteria:

* age from12 to 80 and both sex

Exclusion Criteria:

* patients with other dermatological disorders

Ages: 12 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients with psoriasis
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
the serum level of bioactive lipid mediators in patients with psoriasis | 1 month
  Bioactive lipid mediators (LMs) are potent compounds reported to play a role in the development and resolution of inflammation.

REFERENCES:
- [Background] Sorokin AV, Domenichiello AF, Dey AK, Yuan ZX, Goyal A, Rose SM, Playford MP, Ramsden CE, Mehta NN. Bioactive Lipid Mediator Profiles in Human Psoriasis Skin and Blood. J Invest Dermatol. 2018 Jul;138(7):1518-1528. doi: 10.1016/j.jid.2018.02.003. Epub 2018 Feb 15. PMID 29454560
- [Background] Bakry OA, El Hefnawy S, Mariee AH, El Gendy Y. Urinary Biopyrrins: A New Marker of Oxidative Stress in Psoriasis. Indian J Dermatol. 2016 Mar-Apr;61(2):169-73. doi: 10.4103/0019-5154.177756. PMID 27057016